# STUDY PROTOCOL & STATISTICAL ANALYSIS PLAN

| Official Title: | HYPERTHERMIA AS AN ADDITIONAL TREATMENT<br>FOR THE BIOLOGY AND EXPERIENCE OF<br>DEPRESSION: THE HEATBED STUDY |
|---|---|
| Clinicaltrials.gov # | NCT05041361 |
| Date | 8 April 2024 |
| <b>Development Phase:</b> | Feasibility & Acceptability |
| Sponsor: | Ashley E. Mason, PhD & Frederick M. Hecht, MD UCSF Osher Center for Integrative Health School of Medicine 1545 Divisadero Street Suite 301 San Francisco CA 94115 |
| Principal Investigator: | Name: Ashley E. Mason, PhD<br>E-mail: Ashley.Mason@ucsf.edu |
| Co-Principal | Name: Frederick M. Hecht, MD |
| Investigator | E-mail: Rick.Hecht@ucsf.edu |
| Medical Monitor: | Name: Frederick M. Hecht, MD |
| | E-mail: Rick.Hecht@ucsf.edu |

#### BACKGROUND

Depression recovery is not uniformly linear; people who recover from depression often experience acute improvements, termed 'sudden gains,' early in treatment. Data suggest that participants with clinical depression who receive whole body heating (Hanusch et al., 2013; Janssen et al., 2016) and participants who receive cognitive behavioral therapy (CBT) treatment (Aderka et al., 2012; Tang et al., 1999) show sudden gains. Ascertaining if a treatment comprising both sauna sessions and CBT sessions is feasible and tolerable will allow for further research of this integrative mind-body treatment as a potentially effective and disseminable treatment for clinical depression.

Prior work has demonstrated that whole body heating to an internal temperature of 38.5 °C (101.3 °F) using a head out infrared heating device is tolerable by healthy adults and is associated with significant reductions in clinical depression (Hanusch et al., 2013; Janssen et al., 2016) that characterize sudden gains. This prior work administered a single sauna session in a Heckel heating device, a medical hyperthermia device, and reported improvements in depression symptoms within 1 week of this session. This prior work did not ascertain if additional sauna sessions led to further decreases in depression; a dose-escalation study has not yet been performed. Our earlier pilot project established (in *N*=25 participants) that a readily accessible, commercially available sauna, which the UCSF IRB granted NSR designation, can achieve a core temperature of 101.3 °F without serious adverse events.

In addition to the body-based approach of using sauna as a possible treatment for depression symptoms, we will provide the current gold standard psychotherapy intervention, cognitive behavioral therapy (CBT) to participants. Cognitive behavioral therapy (CBT) is an efficacious, highly disseminable evidence-based treatment for depression. Many therapy modalities can elicit sudden gains; however, sudden gains in cognitive behavioral therapy (CBT) are more frequent and durable than those observed in non-CBT therapies (Aderka et al., 2012). Meta-analytic data suggest that the effects of sudden gains on depression symptoms in the context of CBT treatment are larger (Hedges's g=0.74) and longer lasting than those occurring in the context of non-CBT treatment (Hedges's g=0.23; Aderka et al., 2012). The conceptual framework of sudden gains suggests that such gains can lead to cognitive changes that then lead to further symptom reduction, sparking a positive feedback loop termed an "upward spiral" (Tang & DeRubeis, 1999). Sudden gains in CBT generally follow from "critical" therapy sessions characterized by substantial cognitive change. CBT is an effective manualized psychotherapy that a diverse range of mental health clinicians, including marriage and family therapists (MFTs) and clinical social workers (CSWs), can provide. In many areas, MFTs and CSWs are more readily available and affordable than clinical psychologists. Hence, optimizing an intervention that includes a psychotherapy modality that a range of mental health clinicians can provide strengthens the potential for dissemination.

## References:

Aderka IM, Nickerson A, Bøe HJ, Hofmann SG. Sudden gains during psychological treatments of anxiety and depression: A meta-analysis. *J Consult Clin Psychol*. 2012;80(1):93.

Hanusch, K.-U., Janssen, C. H., Billheimer, D., Jenkins, I., Spurgeon, E., Lowry, C. A., & Raison, C. L. (2013). Whole-body hyperthermia for the treatment of major depression: Associations with thermoregulatory cooling. *American Journal of Psychiatry*, 170(7), 802–804.

Janssen, C. W., Lowry, C. A., Mehl, M. R., Allen, J. J. B., Kelly, K. L., Gartner, D. E., ... Raison, C. L. (2016). Whole-Body Hyperthermia for the Treatment of Major Depressive Disorder: A Randomized Clinical Trial. *JAMA Psychiatry*, 73(8), 789–795.

Tang TZ, DeRubeis RJ. Sudden gains and critical sessions in cognitive-behavioral therapy for depression. *J Consult Clin Psychol*. 1999;67(6):894

| TITLE | EXAMINING THE FEASIBILITY AND ACCEPTABILITY OF SAUNA SESSIONS AND COGNITIVE BEHAVIORAL THERAPY (CBT) FOR PARTICIPANTS WITH CLINICAL DEPRESSION |
|---|---|
| SPONSOR | Ashley E. Mason, PhD |
| CO-SPONSOR | Frederick M. Hecht, MD |
| NUMBER OF<br>SITES | 1 |
| RATIONALE | Depression recovery is not uniformly linear; people who recover from depression often experience acute improvements, termed 'sudden gains,' early in treatment. Data suggest that participants with clinical depression who receive whole body heating (Hanusch et al., 2013; Janssen et al., 2016) and participants who receive cognitive behavioral therapy (CBT) treatment (Aderka et al., 2012; Tang et al., 1999) show sudden gains. Ascertaining if a treatment comprising both sauna sessions and CBT sessions is feasible and tolerable will allow for further research of this integrative mind-body treatment as a potentially effective and disseminable treatment for clinical depression. |
| STUDY DESIGN | Single-arm, unblinded pilot trial |

| PRIMARY<br>OBJECTIVE<br>SECONDARY | Develop a whole-body heating (WBH) + Cognitive Behavioral Therapy (CBT) treatment. We will enroll 16 participants with clinical depression and deliver *4 biweekly WBH (sauna) sessions and 8 weekly CBT sessions. After the first half of enrollment (~n=8) is complete, we will use participant and staff feedback to refine procedures for the remaining enrollment (we will submit any refinements or changes to the treatment to the UCSF IRB approval before implementing them). *Of note, after n=6 participants had completed participation, we reduced the number of WBH sessions from 8 weekly sessions to 4 biweekly (every-other-week) sessions for the remaining 10 participants. To pilot test the feasibility of all assessment procedures in anticipation |
|---|---|
| <b>OBJECTIVES</b> | of a larger trial. |
| NUMBER OF<br>PARTICIPANT<br>S | 16 |
| PARTICIPANT<br>SELECTION<br>CRITERIA | <ul> <li>Inclusion Criteria: <ol> <li>Age of at least 18 years old</li> <li>Current major depressive episode of at least 2 weeks duration as assessed by the Structured Clinical Interview for DSM-5 (SCID) and a Beck Depression Inventory-II (BDI-II) score ≥ 21 at screening</li> <li>Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures</li> <li>Must have smartphone onto which they can download an app from Apple App or Google Play stores</li> <li>Ability to lie supine (on back) for 2 hours (required for sauna sessions)</li> <li>Must be fully vaccinated against COVID-19</li> </ol> </li> <li>Exclusion Criteria: <ol> <li>&gt;30% reduction in BDI-II score between Screen #1 and Screen #2 (conducted ~1 week after Screen #1).</li> <li>Suicide attempt in the past 12 months defined using the SAMHSA suicidality question during the clinician-administered interview or active suicidal ideation as indexed by a score of 3 on the BDI-II suicidality item during the clinician-administered interview.</li> <li>Any of the following medical conditions: cardiovascular disease (other than controlled hypertension), seizure disorder, history of cerebrovascular accident (CVA) or other serious neurological condition (e.g. Parkinson's disease, multiple sclerosis, or dementia), current neoplasia, any active enclosed infection (e.g. dental abscess, joint infection), hemophilia or other cause for</li> </ol> </li> </ul> |

- excessive bleeding (e.g. platelet disorder), or other medical condition that in the opinion of investigators may increase the risk of WBH
- 4. Comorbid psychiatric conditions or history of comorbid psychiatric conditions that might better explain depressive symptoms, including schizophrenia, schizoaffective disorder, Bipolar Disorder I, Obsessive Compulsive Disorder, Anorexia Nervosa, Bulimia Nervosa, Alcohol Dependence, or Drug Dependence
- 5. Known hypersensitivity to hyperthermia and/or infrared exposure
- 6. Inability to fit into the sauna device
- 7. Breast implants
- 8. Pregnancy, active lactation or intention to become pregnant during the study period
- 9. Use of any medication that might impact thermoregulatory capacity, including:
  - diuretics, barbiturates
  - beta-blockers
  - antipsychotic agents
  - anti-cholinergic agents or chronic use of antihistamines
  - aspirin (other than low-dose ASA for prophylactic purposes)
  - medication prescribed for the treatment of depression
     (antidepressant medication [ADM]) including but not
     limited to: selective serotonin reuptake inhibitors [SSRIs],
     Serotonin and norepinephrine reuptake inhibitors [SNRIs],
     Monoamine oxidase inhibitors [MAOIs], Tricyclics
     [TCAs], and atypical antipsychotic and antidepressant
     medications (participants must have been free of these
     medications for at least 4 weeks)
  - antibiotics (past 14 days), pain medication (opioids) due to procedure, e.g., dental procedure (past 14 days), Emergency contraception pill (past 14 days)
  - any other medication that in the judgment of the PI would increase risk of study participation or introduce excessive variance into physiological or behavioral responses to WBH
  - recent use (multiple consecutive doses) of: non-steroidal anti-inflammatory drugs (NSAIDs), systemic corticosteroids, cytokine antagonists
- 10. Regular use of any nicotine products, including cigarettes, vapes, chewing tobacco, or other forms of nicotine (if use is not regular, must be willing to refrain for 24 hours before and 24 hours after sauna session)
- 11. Unwilling to refrain from using marijuana products and alcohol for the 24 hours before and 24 hours after sauna sessions

| | <ul> <li>12. Unwilling to refrain from heavy exercise on the day of sauna sessions</li> <li>13. Unwilling to refrain from engaging with sauna, hot yoga, cold plunges, cryotherapy, and hot tub/jacuzzi outside of study (prospective participant must not have engaged with any of these activities for 30 days prior to their baseline study visit).</li> <li>14. Has begun new psychotherapy treatment in the prior 6 weeks</li> <li>*Note: All medications reported by potential subjects will be reviewed by medical monitor Frederick Hecht, MD. If the medication is determined to not have meaningful impacts on bodily thermoregulatory processes and to not interact with whole body heating, the subject may participate.</li> </ul> |
|---|---|
| TECT | |
| TEST | Portable Sauna Dome – One Person |
| PRODUCT, DOSE, AND | Supine sauna device, head out, body inside of sauna<br>Sauna session approx. 80 – 140 minutes, maximum 140 minutes |
| ROUTE OF | Manufactured by Clearlight Infrared |
| ADMINISTRAT | The state of the s |
| ION | |
| CONTROL PRODUCT, DOSE AND ROUTE OF ADMINISTRAT ION | N/A, all participants receive the same treatment |
| DURATION OF<br>PARTICIPANT<br>PARTICIPATIO<br>N AND | This is a single-center, single-arm, non-randomized experimental study that will include 16 participants. Participants will be in the study for approximately 10 weeks. Total time involved will be approximately ~33.5 hours: |
| DURATION OF<br>STUDY | • E-Screen: Web-based eligibility screen for self-report eligibility criteria o ~10 minutes |
| | <ul> <li>Phone Screen: Phone call to review eligibility, schedule study visits</li> <li>~30 minutes</li> </ul> |
| | <ul> <li>Online Depression Screen: Web-based depression screen</li> <li>~10 minutes</li> </ul> |
| | <ul> <li>In-Person Screen / Baseline Visit: Participant to complete screening procedures, provide informed written consent and receive bill of rights, download Oura Ring app, complete self-report questionnaires and anthropometric assessments</li> <li>~150 minutes</li> </ul> |
| | <ul> <li>Daily depression assessment: Brief web-based surveys assessing depression symptoms each morning</li> <li>~2 minutes each</li> </ul> |

- Sauna Visits 1-4: In-person visits, participant (if female) to complete pregnancy screen if the participant thinks there is a possibility of pregnancy, COVID-19 rapid test, complete questionnaires (all sauna visits), provide blood and saliva samples (Sauna Visits 1, 3 and 4), and complete sauna session
  - $\circ$  ~240-260 minutes each
- Cognitive Behavioral Therapy (CBT) Visits 1-8: In-person visits, participant to receive 50-minute CBT session and complete selfreport measures
  - ~75 minutes each
- Close-out visit: In-person visit, participant to complete questionnaires, complete clinician-administered assessment, provide blood and saliva samples if the participant does not complete a 4th sauna visit, return Oura Ring
  - ~85 minutes

## CONCOMMITA NT MEDICATIONS

### Allowed:

• All medications reported by potential participants will be reviewed by medical monitor Frederick Hecht, MD. If the medication is determined to not have meaningful impacts on bodily thermoregulatory processes and to not interact with whole body heating, the participant may participate.

## Prohibited:

- 1. Use of any medication that might impact thermoregulatory capacity, including: diuretics, barbiturates, beta-blockers, antipsychotic agents, anti-cholinergic agents or chronic use of antihistamines, cytokine antagonists
- 2. Current antidepressant medications (all classes) or use within the past 30 days
- 3. Recent use (multiple consecutive doses) of systemic corticosteroids
- 4. Needing to use antihistamines, aspirin (other than low-dose ASA for prophylactic purposes), non-steroidal anti-inflammatory drugs (NSAIDs), or systemic corticosteroids, on Study Visit days
- 5. Use of any other medication that in the judgment of the PI would increase risk of study participation or introduce excessive variance into physiological or behavioral responses to WBH
- 6. Regular use of any nicotine products, including cigarettes, vapes, chewing tobacco, or other forms of nicotine
- 7. The following medications in these timeframes: Antibiotics (past 14 days), Pain medication (opioids) due to procedure, e.g., dental procedure (past 14 days), Emergency contraception pill (past 14 days)

| EFFICACY<br>EVALUATIONS | See below for primary and secondary endpoints. |
|---|---|
| PRIMARY<br>ENDPOINT | Primary outcomes. The primary endpoint is the average number of planned WBH sessions completed. We have selected this as the primary outcome because prior studies have not assessed the acceptability of multiple sauna sessions and we believe it is important to verify acceptability of multiple sauna sessions before including it in further steps. |
| SECONDARY<br>ENDPOINTS | Secondary outcomes. The secondary endpoints are the average number of planned BDI-II assessments completed and the change in the BDI-II from baseline to the final assessments (12 weeks). |
| OTHER<br>EVALUATIONS | N/A |
| SAFETY<br>EVALUATIONS | Incidence of unexpected adverse events. We will monitor participants for unexpected adverse events and serious adverse events during and following the sauna sessions. |
| PLANNED<br>INTERIM<br>ANALYSES | Due to the current study design and safety profile of this test product (portable sauna dome – one person) and cognitive behavioral therapy (CBT; a standard depression psychotherapy treatment), we do not plan any interim analyses. |
| STATISTICS<br>Primary Analysis<br>Plan | Primary outcome: We initially planned to quantify the number of planned WBH sessions completed and provide this information as the mean number of sessions with the corresponding standard deviation. Because, with Sponsor oversight and permission, we changed the number WBH sessions offered from 8 WBH sessions to 4 WBH sessions to optimize feasibility midway through enrollment, we analyzed the primary outcome separately for participants offered 8 WBH sessions and participants offered 4 WBH sessions. |
| | Secondary outcome: We quantified the number of BDI-II assessments completed and provide this information as the mean number of assessments completed with the corresponding standard deviation. All participants were administered 10 BDI-II assessments. |
| | Secondary outcome: We calculated the change in BDI-II scores from the baseline BDI-II assessment to the final BDI-II assessment (12 weeks) by computing a paired t-test using the final assessment and the baseline assessment, and provide 95% confidence intervals around the mean difference. All participants who completed participation were administered the baseline and final BDI-II assessments. |
| Rationale for<br>Number of<br>Participants | This study (which is funded by NIH/NCCIH and gift funding) will recruit 16 participants and aims to assess feasibility and acceptability of the planned sauna + CBT treatment. We are not aiming to test efficacy in these studies as we do not have adequate sample size. If 14 of 16 participants complete at least 80% of their assigned WBH sessions (87.5%), the 95% CI for this rate will be 71% to 100% (normal approximation to the binomial), which we believe will |

| provide adequate precision | on for feasibility testing. |
|----------------------------|-----------------------------|